CLINICAL TRIAL: NCT03028740
Title: AURORA: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Cenicriviroc for the Treatment of Liver Fibrosis in Adult Subjects With Nonalcoholic Steatohepatitis
Brief Title: AURORA: A Study for the Efficacy and Safety of Cenicriviroc (CVC) for the Treatment of Liver Fibrosis in Adults With Nonalcoholic Steatohepatitis (NASH)
Acronym: AURORA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated early due to lack of efficacy based on the results of the planned interim analysis of Part 1 data.
Sponsor: Tobira Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3152-301-002; 2016-004566-26 (EudraCT Number); 1001 (Registry Identifier: Registro Nacional Estudios Clinicos (RNEC))
Record Dates: First submitted 2017-01-13; First posted 2017-01-23 (Estimated); Results first posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2021-11

CONDITIONS: Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — cenicriviroc

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received cenicriviroc placebo-matching, tablet, orally, once daily for up to approximately 40 months.
  Interventions: Drug: Placebo
- Cenicriviroc 150 mg (Experimental): Participants received cenicriviroc, 150 milligrams (mg), tablet, orally, once daily for up to approximately 40 months.
  Interventions: Drug: Cenicriviroc

INTERVENTIONS:
Drug: Placebo — Cenicriviroc placebo-matching, tablet, orally, once daily for up to approximately 40 months.
  Arms: Placebo
Drug: Cenicriviroc — Cenicriviroc, 150 mg, tablet, orally, once daily for up to approximately 40 months.
  Other Names: CVC
  Arms: Cenicriviroc 150 mg

SUMMARY:
The AURORA study will be conducted to confirm the efficacy and safety of cenicriviroc (CVC) for the treatment of liver fibrosis in adult participants with NASH.

DETAILED DESCRIPTION:
The AURORA study will be conducted in 2 parts. Part 1 will examine the surrogate endpoint of improvement in fibrosis of at least 1 stage (nonalcoholic steatohepatitis clinical research network [NASH CRN]) and no worsening of steatohepatitis at Month 12. Participants from Part 1 will continue into Part 2 and additional participants will be newly randomized in Part 2 to determine long-term clinical outcomes composed of histopathologic progression to cirrhosis, liver-related clinical outcomes, and all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged between 18-75 years
* Ability to understand and sign a written informed consent form (ICF)
* Histological evidence of NASH based on central reading of the Screening biopsy
* Participants included in Part 1 must have histopathological evidence of Stage 2 or 3 liver fibrosis per the NASH CRN System based on central reading of the Screening biopsy slides. Participants newly randomized in Part 2 must have histological evidence of Stage 3 liver fibrosis per the NASH CRN System, based on central reading of the Screening period biopsy slides. Historical biopsy can be used, provided the criteria listed on Item 3a above are fulfilled.
* Females of childbearing potential and males participating in the study must agree to use at least 2 approved methods of contraception throughout the duration of the study and for 30 days after stopping study drug. Females who are postmenopausal must have documentation of cessation of menses for ≥12 months and serum follicle-stimulating hormone (FSH) ≥30 milliunits (mU)/milliliter (mL) at Screening.

Exclusion Criteria:

* Inability to undergo a liver biopsy
* Hepatitis B surface antigen (HBsAg) positive
* Hepatitis C antibody (HCVAb) positive
* Human immunodeficiency virus (HIV)-1 or HIV-2 infection
* Prior or planned liver transplantation
* Other known causes of chronic liver disease
* History or presence of cirrhosis and/or hepatic decompensation including ascites, hepatic encephalopathy or variceal bleeding
* Alcohol consumption greater than 21 units/week for males or 14 units/week for females
* Aspartate transaminase (AST) >200 International units (IU)/liter (L) in males and females at Screening
* Alanine transaminase (ALT) >250 IU/L in males and >200 IU/L in females at Screening
* Hemoglobin A1c (HbA1c) >10% at Screening
* Serum albumin <3.5 gram (g)/deciliter (dL) at Screening
* Estimated glomerular filtration rate (eGFR) < 50 mL/minute (min)/1.73 meter (m)^2 according to the Modification of Diet in Renal Disease (MDRD) equation
* Platelet count <100,000/millimeter (mm)^3
* Total bilirubin >1.5 milligram (mg)/dL
* International normalized ratio (INR) >1.3
* Model of end stage liver disease (MELD) score >12
* Weight reduction, defined as ≥7% of body weight, through bariatric surgery in the past 5 years or bariatric surgery planned during the conduct of the study (including gastric banding and sleeve surgery)
* History of malignancy within the past 5 years or ongoing malignancy other than basal cell carcinoma, or resected noninvasive cutaneous squamous cell carcinoma
* Active, serious infections that require parenteral antibiotic or antifungal therapy within 30 days prior to Screening Visit
* Clinically significant cardiovascular or cerebrovascular disease within the past 3 months
* Females who are pregnant or breastfeeding
* Current or anticipated treatment with radiation therapy, cytotoxic chemotherapeutic agents and immunomodulating agents (eg, interleukins, interferons, cyclosporine, tacrolimus) except for vaccines or short-term corticosteroids
* Receiving a glucagon-like peptide 1 (GLP-1) receptor agonist, a dipeptidyl peptidase 4 (DPP-4) inhibitor, a sodium-glucose cotransporter 2 (SGLT2) and/or sodium-glucose cotransporter (SGLT1) inhibitor, or a thiazolidinedione (TZD) for less than 6 months prior to the Screening period liver biopsy. Participants on a stable therapy with a GLP-1 receptor agonist, DPP-4 inhibitor, SGLT1 and/or SGLT2 inhibitor, or a TZD for at least 6 months prior to the Screening liver biopsy may be considered eligible. (Important Note: if a historical biopsy is to be used, participants need to be on stable therapy for at least 6 months prior to the day historical liver biopsy was performed).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1778 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Rodriguez, Study Director — Allergan
Locations (345):
- United States (203):
  - Summit Internal Medicine, Birmingham, Alabama
  - Cullman Clinical Trials, Cullman, Alabama
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Objective GI D/B/A North Alabama GI Research Center, Madison, Alabama
  - The Institute for Liver Health, Chandler, Arizona
  - Adobe Gastroenterology Research, LLC, Tucson, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Del Sol Research Management LLC, Tucson, Arizona
  - Arkansas Diagnostic Center, Little Rock, Arkansas
  - Franco Felizarta MD, Bakersfield, California
  - Hope Clinical Research, Canoga Park, California
  - GW Research, Chula Vista, California
  - eStudySite, Chula Vista, California
  - Southern California Research Center, Coronado, California
  - Citrus Valley Gastroenterology, Covina, California
  - TriWest Research Associates, El Cajon, California
  - University of San Francisco, Fresno Medical Education Program, Fresno, California
  - Fresno Clinical Research Center (FCRC), Fresno, California
  - National Research Institute, Huntington Park, California
  - University of California San Diego, La Jolla, California
  - eStudySite, La Mesa, California
  - Om Research, Lancaster, California
  - Southern California Kaiser Permanente, Los Angeles Medical Center, Los Angeles, California
  - GastroIntestinal Biosciences, Los Angeles, California
  - Global Research Institute, Los Angeles, California
  - Ruane Medical and Liver Health Institute, Los Angeles, California
  - Cedars-Sinai Medical Group, Los Angeles, California
  - National Research Institute, Los Angeles, California
  - United Medical Doctors, Murrieta, California
  - Palmtree Clinical Research Inc., Palm Springs, California
  - National Research Institute, Panorama City, California
  - Pasadena Liver Center, Pasadena, California
  - Alliance Clinical Research LLC, Poway, California
  - Stanford School of Medicine, Center for Clinical Sciences Research, Redwood City, California
  - Inland Empire Liver Foundation, Rialto, California
  - Precision Research Institute, San Diego, California
  - Southern California Permanente Medical Group, San Diego, California
  - UCSF School of Medicine, San Francisco, California
  - Upland Clinical Research, Upland, California
  - Island View GI, Ventura, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - South Denver Gastroenterology, PC, Englewood, Colorado
  - Western States Clinical Research, Inc., Wheat Ridge, Colorado
  - Gastroenterology Associates of Fairfield County, Bridgeport, Connecticut
  - Yale University - New Haven, New Haven, Connecticut
  - Innovative Medical Research of South Florida, Inc., Aventura, Florida
  - Gastro Florida, Clearwater, Florida
  - Hi Tech and Global Research, LLC, Coral Gables, Florida
  - Top Medical Research, Inc, Cutler Bay, Florida
  - ICR Sites, Doral, Florida
  - Qway Research, LLC, Hialeah, Florida
  - Gastroenterology Associates - Crystal River, Inverness, Florida
  - Mayo Clinic College of Medicine, Jacksonville, Florida
  - Meridien Research, Lakeland, Florida
  - Florida Digestive Health Specialists, Lakewood Rch, Florida
  - Meridien Research, Maitland, Florida
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Bruce W. Carter Department of Veterans Affairs Medical Center, Miami, Florida
  - Optimus U Corporation, Miami, Florida
  - University of Miami Hospital, Miami, Florida
  - Sanchez Clinical Research, Inc, Miami, Florida
  - Genoma Research Group Inc., Miami, Florida
  - Medical Professional Clinical Research Center, INC, Miami, Florida
  - ProLive Medical Research, Miami, Florida
  - San Marcus Research Clinic, Miami Lakes, Florida
  - Advanced Research Institute, Inc., New Port Richey, Florida
  - Bioclinical Research Alliance, Orlando, Florida
  - Omega Research Maitland, LLC, Orlando, Florida
  - IMIC, Inc, Palmetto Bay, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - Gastroenterology Associates of Pensacola, Pensacola, Florida
  - Advanced Medical Research, Port Orange, Florida
  - Tampa General Hospital, Tampa, Florida
  - Guardian Angel Research Center, Tampa, Florida
  - Bioclinica Research, The Villages, Florida
  - Florida Medical Clinic, Zephyrhills, Florida
  - Summit Clinical Research, LLC, Athens, Georgia
  - Digestive Healthcare of Georgia - Atlanta, Atlanta, Georgia
  - Piedmont Healthcare INC., Atlanta, Georgia
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - GI Specialists of Georgia - Marietta Office, Marietta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Investigators Research Group, LLC, Brownsburg, Indiana
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - Aquiant Research, New Albany, Indiana
  - Digestive Research Alliance of Michiana, South Bend, Indiana
  - Iowa Digestive Disease Center, Clive, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kansas Medical Clinic-Gastroenterology, Topeka, Kansas
  - Delta Research Partners, LLC, Bastrop, Louisiana
  - Avant Research Associates LLC, Crowley, Louisiana
  - C-1 Headlands, Inc., Lake Charles, Louisiana
  - Tandem Clinical Research, Marrero, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Nola Research Works, LLC, New Orleans, Louisiana
  - Louisiana Research Center, Shreveport, Louisiana
  - Clinical Trials of America LLC, West Monroe, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Digestive Disease Associates, Catonsville, Maryland
  - Gastro Center of Maryland, Columbia, Maryland
  - Woodholme Gastroenterology Associates, Glen Burnie, Maryland
  - Victory Clinical Research, Greenbelt, Maryland
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Umass Memorial Medical Center, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Minnesota Gastroenterology, P.A., Maplewood, Minnesota
  - National Diabetes and Obesity Research Institute, Biloxi, Mississippi
  - GastroIntestinal Associates, Flowood, Mississippi
  - Clinical Research Professionals, Chesterfield, Missouri
  - Saint Louis University, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Machuca Family Medicine, Las Vegas, Nevada
  - Jubilee Clinical Research, Inc., Las Vegas, Nevada
  - Sierra Clinical Research, Las Vegas, Nevada
  - Excel Clinical Research, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hassman Research Institute, Berlin, New Jersey
  - Amici Clinical Research, Raritan, New Jersey
  - Beth Israel Medical Center, New York, New York
  - NYU Langone Health - Perlmutter Cancer Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Tandem Clinical Research, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Investigational Drug Service, The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Northeast GI Research Division, Concord, North Carolina
  - Duke University, Durham, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Carolina Research, Greenville, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - The Ohio University - Gastroenterology, Hepatology, Columbus, Ohio
  - Digestive Disease Specialist, Inc., Oklahoma City, Oklahoma
  - Options Health Research, Tulsa, Oklahoma
  - Eastern Pennsylvania Gastroenterology and Liver Specialist, Bethlehem, Pennsylvania
  - UPMC -Center for Liver Diseases, Pittsburgh, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Care Access Research, Pottsville, Pottsville, Pennsylvania
  - Digestive Disease Associates, LTD, Wyomissing, Pennsylvania
  - Partners in Clinical Research, Cumberland, Rhode Island
  - University Medical Group, North Providence, Rhode Island
  - Care Access Research-Warwick, Warwick, Rhode Island
  - Rapid City Medical Center, Rapid City, South Dakota
  - Mount Vernon Clinical Research, Chattanooga, Tennessee
  - Gastro One, Germantown, Tennessee
  - Digestive Health Research, Hermitage, Tennessee
  - East Tennessee Research Institute, Johnson City, Tennessee
  - Digestive Health Research, Lebanon, Tennessee
  - UT-Memphis, Methodist University Hospital, Memphis, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - Methodist Dallas Medical Center, Dallas, Texas
  - Liver Center of Texas, Dallas, Texas
  - Synexus, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - San Antonio Military Medical Center, Fort Sam Houston, Texas
  - Baylor Scott & White All Saints Medical Center - Ft. Worth, Fort Worth, Texas
  - Texas Digestive Disease Consultants - Fort Worth, Fort Worth, Texas
  - Digestive Health Associates of Texas-Rockwall, Garland, Texas
  - Therapeutic Concepts, PA, Houston, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Liver Associates of Texas, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Michael E. DeBakey VA Medical Center (MEDVAMC), Houston, Texas
  - St. Luke's Medical Center, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Centex Studies, Houston, Texas
  - Amir Ali Hassan, MD, PA, Houston, Texas
  - Centex Studies, Inc., McAllen, Texas
  - LinQ Research, LLC, Pearland, Texas
  - Quality Research Inc., San Antonio, Texas
  - American Research Corporation, San Antonio, Texas
  - Clinical Trials of Texas Inc, San Antonio, Texas
  - Diabetes & Glandular Disease Clinic, P.A. (DGD), San Antonio, Texas
  - Endeavor Clinical Trials, LLC, San Antonio, Texas
  - Southern Star Research Institute, LLC SAGACT PLLC., San Antonio, Texas
  - Anson Medicine, San Antonio, Texas
  - Mount Olympus Medical Research, LLC, Sugar Land, Texas
  - Texas Digestive Disease Consultants, Webster, Texas
  - Physician's Research Options, LLC, Draper, Utah
  - Intermountain Medical Center, Murray, Utah
  - Advanced Clinical Research - Center for Digestive Health, Riverton, Utah
  - University of Utah, Salt Lake City, Utah
  - Gastroenterology Associates of Northern Virginia, Fairfax, Virginia
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - Liver Institute of Virginia, Newport News, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - McGuire Veterans Affairs Medical Center, Richmond, Virginia
  - VCU Medical Center, Richmond, Virginia
  - Gastroenterology Consultants of Southwest Virginia Research, Roanoke, Virginia
  - Harborview Medical Center, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - Liver Institute Northwest, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Marshall University Joan C. Edwards School of Medicine, Huntington, West Virginia
- Australia (8):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Saint George Hospital, Kogarah, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Center, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Austria (3):
  - Universitatsklinik far Innere Medizin, Graz, Styria
  - Universitatsklinik far Innere Medizin II, Innsbruck, Tyrol
  - Klinikum Wels-Grieskirchen, Wels, Upper Austria
- Belgium (6):
  - Universitair Ziekenhuis Antwerpen, Edegem, Antwerpen
  - Hôpital Erasme, Brussels, Brussels Capital
  - Algemeen Ziekenhuis Maria Middelares, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen
  - Cliniques Universitaires Saint-Luc, Brussels
  - Centre Hospitalier Chretien CHC, Liège
- Brazil (4):
  - Hospital das Clínicas da Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Faculdade de Medicina de São José do Rio Preto Hospital de Base, São José do Rio Preto, São Paulo
  - Hospital Universitário Clementino Fraga Filho, Rio de Janeiro
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo
- Canada (6):
  - University of Calgary Liver Unit, Calgary, Alberta
  - Bailey Health Clinic, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - William Osler Health Centre, Brampton Memorial Hospital Campus, Brampton, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - Ecogene-21, Chicoutimi, Quebec
- Centro de Investigaciones Clínicas Viña del Mar, Viña del Mar, Región de Valparaíso, Chile
- France (14):
  - CHU de Strasbourg, Strasbourg, Alsace
  - CHU De Bordeaux - Hôpital Haût-Lévèque CMC Magellan Unita de Recherche Clinique, Pessac, Aquitaine
  - Centre Hospitalier Universitaire Estaing, Clermont-Ferrand, Aubergne
  - Centre Hospitalier Universitaire Grenoble, Grenoble, Auvergne-Rhône-Alpes
  - Centre Hospitalier Universitaire de Rennes- Hôpital Pontchaillou, Rennes, Brittany Region
  - Centre Hospitalier Regional et Universitaire de Besancon - L'Hopital Jean Minjoz, Besançon, Franche-Comte
  - CHU de Montpellier, Montpellier, Languedoc-Roussillon
  - Centre Hospitalier Universitaire de Rouen CHU de Rouen Hopital Charles-Nicolle, Rouen, Normandy
  - Center Hospitalier Universitaire d'Angers, Angers, Pays de la Loire Region
  - Hapital Sud Service d'Hepato- Gastroentarologie, Amiens, Picardie
  - Centre Hospitalier Universitaire de Nice Hôpital l'Archet, Nice, Provence-Alpes-Côte d'Azur Region
  - Hopital Avicenne, Bobigny
  - Departement d'Hacpatologie, Clichy, Île-de-France Region
  - Hôpital Saint Antoine, Paris, Île-de-France Region
- Germany (13):
  - Synexus Clinical Research GmbH, Prüfzentrum Frankfurt, Frankfurt am Main, Hesse
  - Philipps-Universität und Universitätsklinikum Gießen und Marburg GmbH, Marburg, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Gastroenterologische Gemeinschaftspraxis, Herne, Nordhein-Westfalen
  - Uniklinik RWTH Aachen, Aachen, North Rhine-Westphalia
  - Uniklinik Köln, Cologne, North Rhine-Westphalia
  - Universitätsmedizin der Johannes Gutenberg Universität Mainz, Mainz, Rhineland-Palatinate
  - Universitätsklinikum des Saarlandes, Homburg, Saarland
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Praxis Driesener Strasse, Berlin
  - Synexus Clinical Research GmbH, Prüfzentrum Berlin, Berlin
  - Charité Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
- Greece (2):
  - Thomopoulos Gastroenterology Dept., Patra, Peloponnese
  - Hippokratio Hospital, Thessaloniki
- Hong Kong (2):
  - Prince of Wales Hospital, Shatin, New Territories
  - Alice Ho Miu Ling Nethersole Hospital, Shatin, New Territories
- Hungary (3):
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár, Somogy County
  - SYNEXUS Magyarország Kft. - Budapest DRS, Budapest
  - Synexus Magyarorszag Egeszsegugyi Szolgaltato Kft, Debrecen
- Israel (9):
  - EMMS MC, Nazareth, Jerusalem
  - Rambam Health Care Campus - Rambam Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Institute of Gastroenterology and Liver Diseases, Jerusalem
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center Beilinson Hospital, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
- Italy (8):
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, Milano
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Azienda Ospedaliera Universitaria Careggi SOD Medicina Interna ed Epatologia, Florence
  - ASST Santi Paolo e Carlo, Milan
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone, Palermo
  - Fondazione Policlinico Tor Vergata, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Mexico (4):
  - Consultorio Médico Dr. Alma Laura Ladron de Guevara, Mexico City, Mexico City
  - JM Research - Cuernavaca, Cuernavaca, Morelos
  - Investigaciones Medicas Cisneros, Monterrey, Nuevo León
  - Consultorio Dra. Maria Sarai Gonzalez Huezo, Metepec
- New Zealand (2):
  - Auckland City Hospital, Grafton, Auckland
  - Middlemore Clinical Trials, Papatoetoe, Auckland
- Oslo Universitetssykehus-Ullevål, Oslo, Norway
- Poland (13):
  - Centrum Badan Klinicznych Piotr Napora Lekarze Spólka Partnerska, Wroclaw, Lower Silesian Voivodeship
  - EMC Instytut Medyczny, Wroclaw, Lower Silesian Voivodeship
  - Szpital Specjalistyczny Nr 1 w Bytomiu, Bytom, Silesian Voivodeship
  - ID Clinic Arkadiusz Pisula, Mysłowice, Silesian Voivodeship
  - Synexus Polska Sp z o o Oddzial w Poznaniu, Poznan, Wielkopolska
  - Synexus Polska Sp. z o.o. Oddzial we Wroclawiu, Wroclaw, Wroclaw
  - Synexus Polska Sp. Z o.o. Oddzial w Czestochowie, Częstochowa
  - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gdansk
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni ul., Gdynia
  - Synexus SCM Sp. z o.o. Oddzial, Katowice
  - Synexus Polska Sp. z o.o. Oddział w Warszawie, Warsaw
  - Synexus Polska Sp. z o.o. Oddział w Łodzi, Lodz, Łódź Voivodeship
  - Wojewódzki Specjalistyczny Szpital im. dr Wl. Bieganskiego w Lodzi, Lódz, Łódź Voivodeship
- Portugal (2):
  - Presa-Ramos, Vila Real, Lordelo
  - Unidade Local de Saúde do Alto Minho, Viana do Castelo
- Puerto Rico (2):
  - Clinical Research Puerto Rico, San Juan, PR
  - Fundacion de Investigacion De Diego, San Juan
- Institutul Regional de Gastroenterologie si Hepatologie Prof. Dr. O Fodor, Cluj-Napoca, Cluj, Romania
- Russia (3):
  - Clinic Professor Gorbakova, Krasnogorsk, Moscow
  - Sklifosovsky Scientific Research Institution of Emergency Care, Moscow
  - Moscow Regional Research and Clinical Institute M.F. Vladimirsky, Moscow
- National University Hospital, Singapore, Singapore
- Spain (13):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Donostia, Donostia / San Sebastian, Guipuzcoa
  - Complejo Hospitalario Torrecardenas, Almería
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Ramón Y Cajal, Madrid
  - Hospital Clínico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Nuestra Senora de Valme, Seville
  - Consorci Hospital General Universitari de València, Valencia
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Switzerland (2):
  - Kantonsspital St.Gallen Klinik für, Sankt Gallen, Canton of St. Gallen
  - Universitaetsspital Bern Inselspital, Bern
- Taiwan (3):
  - Chia-Yi Christian Hospital, Chiayi City, Chiayi
  - China Medical University Hospital, Taichung, Taichung City
  - Chang Gung Medical Foundation-LinKou Branch, Taoyuan District
- United Kingdom (15):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, England
  - Hull and East Yorkshire Hospitals NHS Trust, Hull, England
  - Royal Free London NHS Foundation Trust, London, England
  - Kings College Hospital NHS Foundation Trust, London, England
  - Chelsea and Westminster Hospital NHS Foundation Trust, London, England
  - Luton and Dunstable Hospital NHS Foundation Trust, Luton, England
  - Newcastle Upon the Tyne Hospitals, Newcastle, England
  - Nottingham Digestive Diseases Biomedical Research Unit, Nottingham, England
  - Plymouth Hospitals NHS Trust, Plymouth, England
  - Royal Stoke University Hospital, Stoke-on-Trent, England
  - St James's University Hospital, Leeds, West Yorkshire
  - Synexus Hexham Clinical Research Centre, Hexham
  - Synexus Lancashire Clinical Research Centre, Lancaster
  - Barts Health NHS Trust The Royal London Hospital, London
  - University Hospital of South Manchester NHS Foundation Trust, Manchester

REFERENCES:
- [Derived] Anstee QM, Neuschwander-Tetri BA, Wai-Sun Wong V, Abdelmalek MF, Rodriguez-Araujo G, Landgren H, Park GS, Bedossa P, Alkhouri N, Tacke F, Sanyal AJ. Cenicriviroc Lacked Efficacy to Treat Liver Fibrosis in Nonalcoholic Steatohepatitis: AURORA Phase III Randomized Study. Clin Gastroenterol Hepatol. 2024 Jan;22(1):124-134.e1. doi: 10.1016/j.cgh.2023.04.003. Epub 2023 Apr 13. PMID 37061109

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1778 participants were randomized into the study, of which 1293 participated in Part 1 of the study. The study was terminated early, and Part 2 did not enroll the planned number of participants. Therefore, the Part 1 and Part 2 data were combined and reported as the Full Study Cohort for reporting of the Part 2 efficacy endpoints and the safety endpoints.
Period: Overall Study
Arm/Group | Placebo | Cenicriviroc 150 mg
Started | 593 | 1185
Full Study Cohort: Received Study Drug | 589 | 1180
Participated in Part 1 | 432 | 861
Part 1: Received Study Drug | 429 | 859
Completed | 0 | 0
Not Completed | 593 | 1185
Not completed — Did not Receive Study Drug | 4 | 5
Not completed — Adverse Event | 8 | 26
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 48 | 101
Not completed — Lost to Follow-up | 30 | 54
Not completed — Physician Decision | 4 | 11
Not completed — Protocol Violation | 4 | 8
Not completed — Non-compliance with Study Drug | 0 | 2
Not completed — Study Terminated by Sponsor | 467 | 917
Not completed — Protocol-specified Withdrawal Criteria Met | 27 | 55
Not completed — Reason not Specified | 1 | 5

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat (mITT) Population for the Full Study Cohort included participants randomly assigned to a treatment group who received at least one dose of study drug in Parts 1 and 2 of the study combined.
Groups:
- Cenicriviroc 150 mg: Participants received cenicriviroc,150 mg, tablet, orally, once daily for up to approximately 40 months.
- Total: Total of all reporting groups
Arm/Group | Placebo | Cenicriviroc 150 mg | Total
Number analyzed (Participants) | 589 | 1180 | 1769
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (11.04) | 55.2 (10.76) | 55.4 (10.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 354 | 749 | 1103
  Male | 235 | 431 | 666
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 172 | 315 | 487
  Not Hispanic or Latino | 417 | 865 | 1282
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 8 | 15
  Asian | 22 | 45 | 67
  Native Hawaiian or Other Pacific Islander | 2 | 7 | 9
  Black or African American | 14 | 38 | 52
  White | 539 | 1075 | 1614
  More than one race | 3 | 6 | 9
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percentage of Participants With Improvement in Fibrosis by at Least 1 Stage and No Worsening of Steatohepatitis on Liver Histology at Month 12
Description: Fibrosis stage was evaluated using the Nonalcoholic Steatohepatitis Clinical Research Network (NASH CRN) Fibrosis Staging System with stages: 0=none; 1=perisinusoidal or periportal; 1A=mild, zone 3, perisinusoidal; 1B=moderate, zone 3, perisinusoidal; 1C=portal/periportal; 2=perisinusoidal and portal/periportal; 3=bridging fibrosis; 4=cirrhosis. No worsening of steatohepatitis was defined as no worsening of lobular inflammation or hepatocellular ballooning grade as per scoring in relevant nonalcoholic fatty liver disease activity score (NAS) categories. NAS is a semiquantitative scoring system based on the unweighted sum of: steatosis (0=<5% to 3=>66%), lobular inflammation (0=no foci to 3=>4 foci/200x), and hepatocellular ballooning (0=none to 2=many cells/prominent ballooning) scores. Improvement in fibrosis is a decrease in the NASH CRN fibrosis stage.
Time Frame: Month 12
Population: mITT Population for Part 1 included participants randomly assigned to a treatment group who received at least one dose of study drug in Part 1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Cenicriviroc 150 mg
Number analyzed (Participants) | 429 | 859
percentage of participants | 25.5 [21.5 to 29.9] | 22.3 [19.6 to 25.2]
Statistical Analysis 1: Comparison: Placebo vs Cenicriviroc 150 mg; Test type: Superiority; p = 0.2067, Cochran-Mantel-Haenszel — P-value was based on Cochran-Mantel-Haenszel general association test comparing Cenicriviroc vs Placebo, controlling for factors (randomization strata: fibrosis stage [2 vs 3] and presence or absence of Type 2 diabetes mellitus (T2DM) at Baseline); Percentage Difference = -3.2, 95% CI 2-sided [-8.2 to 1.9]
Statistical Analysis 2: Comparison: Placebo vs Cenicriviroc 150 mg; Test type: Superiority; Odds Ratio (OR) = 0.8369, 95% CI 2-sided [0.6341 to 1.1044] — Odds Ratio was based on Mantel-Haenszel estimates comparing Cenicriviroc vs Placebo, controlling for factors (randomization strata: fibrosis stage [2 vs 3] and presence or absence of T2DM at Baseline)

2. Primary Outcome: Time to First Occurrence of Adjudicated Events in the Full Study Cohort
Description: Time to first occurrence from Baseline was defined as the number of days from the first dose of randomized investigational product to the onset of the first occurrence of any of the following adjudicated events: death (all cause), histopathologic progression to cirrhosis, liver transplant, model for end stage liver disease (MELD) score ≥15, ascites, hospitalization for onset of: variceal bleed, hepatic encephalopathy, spontaneous bacterial peritonitis. MELD is a scoring system for assessing the severity of chronic liver disease and uses the participant's values for total bilirubin, serum creatinine, and the international normalized ratio for prothrombin time to predict survival. MELD score ranges from 6 (less ill) to 40 (gravely ill) with scores and mortality probability being: Score 40=71.3% mortality; Scores 30-39=52.6% mortality; Scores 20-29=19.6% mortality; Scores10-19=6.0% mortality; Score 9 or less=1.9% mortality.
Time Frame: From first dose of study drug to onset of first occurrence of the event (Up to approximately 42 months)
Population: mITT Population for the full study cohort included participants randomly assigned to a treatment group who received at least one dose of study drug in Parts 1 and 2 of the study combined.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Cenicriviroc 150 mg
Number analyzed (Participants) | 589 | 1180
days | NA [NA to NA] — Median, lower and upper limit of 95% confidence interval (C.I.) were not estimable due to low number of participants with events. | NA [NA to NA] — Median, lower and upper limit of 95% C.I. were not estimable due to low number of participants with events.

3. Secondary Outcome: Part 1: Percentage of Participants With Improvement in Fibrosis by at Least 2 Stages and No Worsening of Steatohepatitis on Liver Histology at Month 12
Description: Fibrosis stage was evaluated using the NASH CRN Fibrosis Staging System with stages: 0=none; 1=perisinusoidal or periportal; 1A=mild, zone 3, perisinusoidal; 1B=moderate, zone 3, perisinusoidal; 1C=portal/periportal; 2=perisinusoidal and portal/periportal; 3=bridging fibrosis; 4=cirrhosis. No worsening of steatohepatitis was defined as no worsening of lobular inflammation or hepatocellular ballooning grade as per scoring in relevant NAS categories. NAS is a semiquantitative scoring system based on the unweighted sum of: steatosis (0=<5% to 3=>66%), lobular inflammation (0=no foci to 3=>4 foci/200x), and hepatocellular ballooning (0=none to 2=many cells/prominent ballooning) scores. Improvement in fibrosis is a decrease in the NASH CRN fibrosis stage.
Time Frame: Month 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Cenicriviroc 150 mg
Number analyzed (Participants) | 429 | 859
percentage of participants | 8.3 [6.0 to 11.3] | 6.6 [5.1 to 8.5]
Statistical Analysis 1: Comparison: Placebo vs Cenicriviroc 150 mg; Test type: Superiority; p = 0.2827, Cochran-Mantel-Haenszel — P-value was based on Cochran-Mantel-Haenszel general association test comparing Cenicriviroc vs Placebo, controlling for factors (randomization strata: fibrosis stage [2 vs 3] and presence or absence of T2DM at Baseline); Percentage Difference = -1.7, 95% CI 2-sided [-4.8 to 1.5]
Statistical Analysis 2: Comparison: Placebo vs Cenicriviroc 150 mg; Test type: Superiority; Odds Ratio (OR) = 0.7844, 95% CI 2-sided [0.5032 to 1.2229] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Part 1: Percentage of Participants With Improvement in Fibrosis by at Least 1 Stage Regardless of Effect on Steatohepatitis at Month 12
Description: Fibrosis stage was evaluated using the NASH CRN Fibrosis Staging System with stages 0=none, 1=perisinusoidal or periportal, 1A=mild, zone 3, perisinusoidal, 1B=moderate, zone 3, perisinusoidal, 1C=portal/periportal, 2=perisinusoidal and portal/periportal, 3=bridging fibrosis, 4=cirrhosis.
Time Frame: Month 12
Population: mITT Population for Part 1 included participants randomly assigned to a treatment group who received at least one dose of study drug in Part 1. Overall number analyzed is the number of participants with data available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cenicriviroc 150 mg: Participants received cenicriviroc, 150 mg, tablet, orally, once daily for up to approximately 40 months.
Arm/Group | Placebo | Cenicriviroc 150 mg
Number analyzed (Participants) | 348 | 692
percentage of participants | 33.3 [28.6 to 38.4] | 30.6 [27.3 to 34.2]
Statistical Analysis 1: Comparison: Placebo vs Cenicriviroc 150 mg; Test type: Superiority; p = 0.4054, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Percentage Difference = -2.7, 95% CI 2-sided [-8.7 to 3.3]
Statistical Analysis 2: Comparison: Placebo vs Cenicriviroc 150 mg; Test type: Superiority; Odds Ratio (OR) = 0.8877, 95% CI 2-sided [0.6709 to 1.1744] — [estimate comment as in outcome 1, analysis 2]

5. Secondary Outcome: Part 1: Percentage of Participants With Improvement in Fibrosis by at Least 2 Stages Regardless of Effect on Steatohepatitis at Month 12
Description: as for outcome 4
Time Frame: Month 12
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Cenicriviroc 150 mg
Number analyzed (Participants) | 348 | 692
percentage of participants | 10.3 | 8.8

6. Secondary Outcome: Percentage of Participants With Improvement in Fibrosis by at Least 1 Stage and No Worsening of Steatohepatitis on Liver Biopsy at Month 12 in the Full Study Cohort
Description: as for outcome 3
Time Frame: Month 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Cenicriviroc 150 mg
Number analyzed (Participants) | 589 | 1180
percentage of participants | 25.0 [21.2 to 29.2] | 22.0 [19.4 to 24.8]

7. Secondary Outcome: Percentage of Participants With Improvement in Fibrosis by at Least 1 Stage Regardless of Effect on Steatohepatitis on Liver Biopsy at Month 12 in the Full Study Cohort
Description: as for outcome 4
Time Frame: Month 12
Population: mITT Population for the full study cohort included participants randomly assigned to a treatment group who received at least one dose of study drug in Parts 1 and 2 of the study combined. Overall number analyzed is the number of participants with data available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Drug: Placebo: Participants received cenicriviroc placebo-matching, tablet, orally, once daily for up to approximately 40 months.
- Drug: Cenicriviroc 150 mg: Participants received cenicriviroc, 150 mg, tablet, orally, once daily for up to approximately 40 months.
Arm/Group | Drug: Placebo | Drug: Cenicriviroc 150 mg
Number analyzed (Participants) | 373 | 741
percentage of participants | 33.2 [28.7 to 38.2] | 30.5 [27.3 to 33.9]

8. Secondary Outcome: Percentage of Participants With Improvement in Fibrosis by at Least 2 Stages and No Worsening of Steatohepatitis on Liver Biopsy at Month 12 in the Full Study Cohort
Description: as for outcome 3
Time Frame: Month 12
Population: mITT Population for the full study cohort included participants randomly assigned to a treatment group who received at least one dose of study drug for Parts 1 and 2 of the study combined.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Cenicriviroc 150 mg
Number analyzed (Participants) | 589 | 1180
percentage of participants | 8.3 [5.9 to 11.1] | 6.8 [5.2 to 8.6]

9. Secondary Outcome: Percentage of Participants With Improvement in Fibrosis by at Least 2 Stages Regardless of Effect on Steatohepatitis on Liver Biopsy at Month 12 in the Full Study Cohort
Description: as for outcome 4
Time Frame: Month 12
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Cenicriviroc 150 mg
Number analyzed (Participants) | 373 | 741
percentage of participants | 9.9 | 8.9

10. Secondary Outcome: Percentage of Participants With Improvement in Fibrosis by at Least 1 Stage and No Worsening of Steatohepatitis on Liver Biopsy at Month 60 in the Full Study Cohort
Description: as for outcome 3
Time Frame: Month 60
Population: No data was collected as the study was terminated and no participants reached the Month 60 timepoint.
Arm/Group | Placebo | Cenicriviroc 150 mg
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Percentage of Participants With Improvement in Fibrosis by at Least 1 Stage Regardless of Effect on Steatohepatitis on Liver Biopsy at Month 60 in the Full Study Cohort
Description: as for outcome 4
Time Frame: Month 60
Population: No data was collected as the study was terminated and no participants reached the Month 60 timepoint.
Arm/Group | Placebo | Cenicriviroc 150 mg
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Percentage of Participants With Improvement in Fibrosis by at Least 2 Stages and No Worsening of Steatohepatitis on Liver Biopsy at Month 60 in the Full Study Cohort
Description: as for outcome 3
Time Frame: Month 60
Population: No data was collected as the study was terminated and no participants reached the Month 60 timepoint.
Arm/Group | Placebo | Cenicriviroc 150 mg
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Percentage of Participants With Improvement in Fibrosis by at Least 2 Stages Regardless of Effect on Steatohepatitis on Liver Biopsy at Month 60 in the Full Study Cohort
Description: Fibrosis stage was evaluated using NASH CRN Fibrosis Staging System with stages 0=None, 1=Perisinusoidal or periportal, 1A=Mild, zone 3, perisinusoidal, 1B=Moderate, zone 3, perisinusoidal, 1C=Portal/periportal, 2=Perisinusoidal and portal/periportal, 3=Bridging fibrosis, 4=Cirrhosis.
Time Frame: Month 60
Population: No data was collected as the study was terminated and no participants reached the Month 60 timepoint.
Arm/Group | Placebo | Cenicriviroc 150 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose through 30 days after the last dose of study drug (Up to approximately 42 months)
Description: All-cause Mortality: All enrolled participants. Serious Adverse Events and Other Adverse Events: Safety Population for the full study cohort included participants who received at least one dose of study drug in Parts 1 and 2 of the study combined.
Arm/Group | Placebo | Cenicriviroc 150 mg
All-Cause Mortality (participants affected / at risk) | 2/593 | 6/1185
Serious Adverse Events (participants affected / at risk) | 70/589 | 159/1180
Other Adverse Events (participants affected / at risk) | 218/589 | 425/1180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=589) | Cenicriviroc 150 mg (N=1180)
Blood loss anaemia (Blood and lymphatic system disorders) | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 4
Coronary artery disease (Cardiac disorders) | 0 | 4
Angina pectoris (Cardiac disorders) | 0 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 3
Myocardial infarction (Cardiac disorders) | 1 | 2
Acute coronary syndrome (Cardiac disorders) | 0 | 2
Aortic valve incompetence (Cardiac disorders) | 0 | 2
Aortic valve disease (Cardiac disorders) | 0 | 1
Aortic valve disease mixed (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Pulseless electrical activity (Cardiac disorders) | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 0/235 | 1/431 — Number of participants at risk in each arm is based on the male population.
Vertigo (Ear and labyrinth disorders) | 1 | 4
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Hypoparathyroidism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Thyroid mass (Endocrine disorders) | 1 | 0
Visual impairment (Eye disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 2 | 6
Colitis (Gastrointestinal disorders) | 1 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Mesenteric panniculitis (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 4
Fatigue (General disorders) | 0 | 2
Chest pain (General disorders) | 1 | 1
Death (General disorders) | 0 | 1
Generalised oedema (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 2 | 6
Pneumonia (Infections and infestations) | 4 | 5
COVID-19 (Infections and infestations) | 2 | 5
Cellulitis (Infections and infestations) | 2 | 4
Sepsis (Infections and infestations) | 5 | 2
Diverticulitis (Infections and infestations) | 2 | 2
Gastroenteritis (Infections and infestations) | 2 | 1
Pyelonephritis (Infections and infestations) | 2 | 1
Osteomyelitis (Infections and infestations) | 1 | 1
Acute sinusitis (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Gallbladder empyema (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 1
Postoperative abscess (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Herpes zoster oticus (Infections and infestations) | 1 | 0
Perineal abscess (Infections and infestations) | 1 | 0
Vulval cellulitis (Infections and infestations) | 1/354 | 0/749 — Number of participants at risk in each arm is based on the female population.
Fall (Injury, poisoning and procedural complications) | 5 | 2
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 | 2
Procedural pain (Injury, poisoning and procedural complications) | 1 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 2
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Post procedural contusion (Injury, poisoning and procedural complications) | 0 | 1
Post procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 3 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Snake bite (Injury, poisoning and procedural complications) | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 1
Serum ferritin increased (Investigations) | 0 | 1
Blood uric acid increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Alkalosis hypochloraemic (Metabolism and nutrition disorders) | 0 | 1
Alkalosis hypokalaemic (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 2
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/235 | 2/431 — Number of participants at risk in each arm is based on the male population.
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/354 | 1/749 — Number of participants at risk in each arm is based on the female population.
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma of eyelid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/354 | 0/749 — Number of participants at risk in each arm is based on the female population.
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 3
Transient ischaemic attack (Nervous system disorders) | 1 | 3
Paraesthesia (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 1 | 1
Loss of consciousness (Nervous system disorders) | 1 | 1
Brain stem infarction (Nervous system disorders) | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Radial nerve palsy (Nervous system disorders) | 0 | 1
Coma (Nervous system disorders) | 1 | 0
Hypersomnia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/354 | 0/749 — Number of participants at risk in each arm is based on the female population.
Device dislocation (Product Issues) | 0 | 1
Depression (Psychiatric disorders) | 1 | 2
Suicidal ideation (Psychiatric disorders) | 1 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Psychiatric decompensation (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 4
Acute kidney injury (Renal and urinary disorders) | 1 | 3
Haematuria (Renal and urinary disorders) | 0 | 2
Renal colic (Renal and urinary disorders) | 0 | 2
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/235 | 1/431 — Number of participants at risk in each arm is based on the male population.
Metrorrhagia (Reproductive system and breast disorders) | 0/354 | 1/749 — Number of participants at risk in each arm is based on the female population.
Polycystic ovaries (Reproductive system and breast disorders) | 0/354 | 1/749 — Number of participants at risk in each arm is based on the female population.
Endometrial hyperplasia (Reproductive system and breast disorders) | 1/354 | 0/749 — Number of participants at risk in each arm is based on the female population.
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Phlebolith (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=589) | Cenicriviroc 150 mg (N=1180)
Nausea (Gastrointestinal disorders) | 39 | 104
Diarrhoea (Gastrointestinal disorders) | 56 | 92
Abdominal pain upper (Gastrointestinal disorders) | 26 | 64
Abdominal pain (Gastrointestinal disorders) | 30 | 56
Fatigue (General disorders) | 33 | 74
Urinary tract infection (Infections and infestations) | 33 | 57
Upper respiratory tract infection (Infections and infestations) | 39 | 41
Arthralgia (Musculoskeletal and connective tissue disorders) | 35 | 68
Back pain (Musculoskeletal and connective tissue disorders) | 36 | 54
Headache (Nervous system disorders) | 30 | 64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT03028740/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT03028740/SAP_001.pdf